CLINICAL TRIAL: NCT05293873
Title: Outcomes of Autologous Bone Marrow-derived Mononuclear Cell Transplantation in the Management of Neurological Sequelae After Traumatic Brain Injury
Brief Title: Outcomes of Autologous Bone Marrow-derived Mononuclear Cell Transplantation in the Management of Neurological Sequelae
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VinmecISC1805
Record Dates: First submitted 2019-03-27; First posted 2022-03-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sequelae of Injuries of Head
Keywords: traumatic brain injury; mononuclear cell; neurological sequelae
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (BM-MNC trasnplatation) (Experimental): Autologous bone marrow-derived mononuclear cell will transplant at baseline, and the second transplantation will be performed 6 months after the first transplantation and combination with rehabilitation therapy
  Interventions: Biological: autologous bone marrow-derived mononuclear cell transplantation; Other: Rehabilitation therapy
- Control group (Other): rehabilitation therapy
  Interventions: Other: Rehabilitation therapy

INTERVENTIONS:
Biological: autologous bone marrow-derived mononuclear cell transplantation — Bm-MNC will be transplanted at baseline, and the second transplantation will be performed 6 months after the first transplantation
  Arms: Treatment (BM-MNC trasnplatation)
Other: Rehabilitation therapy — Rehabilitation therapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous bone marrow-derived mononuclear cell transplantation in the management of neurological sequelae after traumatic brain injury

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of autologous bone marrow-derived mononuclear cell transplantation in 25 patients with neurological sequelae after traumatic brain injury compared with 25 patients in control group (no intervention) at the time points of baseline, 3rd month (D90), 6th month (D180), and 12th month (D360).

ELIGIBILITY:
Inclusion Criteria:

* Age: from 20 to 50 years
* Gender: either sex
* Duration after Brain trauma: 6 - 12 months
* Functional Independence Measure - FIM < 69
* Closed head injury

Exclusion Criteria:

* Neurologic impairment or neurological disease before the time of the accident.
* Active infections
* Tumours or failure of heart, lung, liver or kidney, respiratory distress syndrome
* Anaemia, clotting disorder
* Cancer
* Pregnancy
* Alcoholic
* Patient was unemployed or did not attend school before the accident.
* Severe injuries: spinal cord injury, pelvic inflammation, cardiopulmonary

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events | up to the 12-month period following treatment
  Incidence of the adverse events or serious adverse events after transplantation
Functional Independence Measure | up to the 12-month period following treatment
  Functional Independence Measure assess and grade the functional status of patient
Extended Glasgow Outcome Scale | up to the 12-month period following treatment
  Extended Glasgow Outcome Scale classifies global outcome in TBI survivors

SECONDARY OUTCOMES:
Short Form 36 | up to the 12-month period following treatment
  Short Form 36 items will be performed to evaluate the overall health of the patients for their quality of life
to monitor the functional metabolic changes in the brain of the patients | up to the 12 months after transplantation
  The PET-CT scan will be repeated to monitor the functional metabolic changes in the brain of the patients

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen TL, Nguyen HP, Nguyen TK. The effects of bone marrow mononuclear cell transplantation on the quality of life of children with cerebral palsy. Health Qual Life Outcomes. 2018 Aug 14;16(1):164. doi: 10.1186/s12955-018-0992-x. PMID 30107811
- [Background] Nguyen LT, Nguyen AT, Vu CD, Ngo DV, Bui AV. Outcomes of autologous bone marrow mononuclear cells for cerebral palsy: an open label uncontrolled clinical trial. BMC Pediatr. 2017 Apr 12;17(1):104. doi: 10.1186/s12887-017-0859-z. PMID 28403842
- [Background] Eggenberger S, Boucard C, Schoeberlein A, Guzman R, Limacher A, Surbek D, Mueller M. Stem cell treatment and cerebral palsy: Systemic review and meta-analysis. World J Stem Cells. 2019 Oct 26;11(10):891-903. doi: 10.4252/wjsc.v11.i10.891. PMID 31692977
- [Background] Bansal H, Verma P, Agrawal A, Leon J, Sundell IB, Koka PS. A Short Study Report on Bone Marrow Aspirate Concentrate Cell Therapy in Ten South Asian Indian Patients with Autism. J Stem Cells. 2016;11(1):25-36. PMID 28296862
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477